CLINICAL TRIAL: NCT05808764
Title: A Phase II, Open-label Study to Investigate the Pharmacokinetics and Safety of Risdiplam in Infants With Spinal Muscular Atrophy
Brief Title: A Study to Investigate the Pharmacokinetics and Safety of Risdiplam in Infants With Spinal Muscular Atrophy
Acronym: PUPFISH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN44619; 2023-505602-42-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-30; First posted 2023-04-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Risdiplam (Experimental): Participants will receive risdiplam once daily for 28 days.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — Participants will receive 0.15 mg/kg risdiplam orally once daily for 28 days.
  Other Names: Evrysdi

SUMMARY:
This study will evaluate the pharmacokinetics (PK) and safety of risdiplam in participants with spinal muscular atrophy (SMA) under 20 days of age at first dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female newborn infant aged <20 days at first dose
* Newborn infants with genetic diagnosis of 5q-autosomal recessive SMA or newborn infants identified as positive for SMA via newborn screening or via prenatal testing.
* Gestational age equal to or greater than 37 weeks
* Receiving adequate nutrition and hydration at the time of screening
* Adequately recovered from any acute illness at baseline and considered well enough to participate in the study
* Parent/caregiver is willing to consider nasogastric, nasojejunal, or gastrostomy tube placement during the study to maintain safe hydration, nutrition, and treatment delivery, if recommended by the investigator.

Exclusion Criteria:

* Presence of clinical symptoms or signs consistent with SMA Type 0
* In the opinion of the investigator, inadequate venous or capillary blood access for the study procedures
* Systolic blood pressure or diastolic blood pressure or heart rate abnormalities
* Presence of clinically relevant electrocardiogram (ECG) abnormalities
* The infant (or the person breastfeeding the infant) taking any of the following: any inhibitor of CYP3A4 taken within 2 weeks (or within 5 times the elimination half-life, whichever is longer) prior to dosing, any inducer of CYP3A4 taken within 4 weeks (or within 5 times the elimination half-life, whichever is longer prior to dosing, and/or use of any multidrug and toxin extrusion (MATE) substrates taken within 2 weeks (or within 5 times the elimination half-life, whichever is longer) prior to dosing
* Concurrent or previous administration of nusinersen or onasemnogene abeparvovec
* Clinically significant abnormalities in laboratory test

Max Age: 19 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentrations of Risdiplam | From Day 1 through Day 28
Area Under the Plasma Concentration-Time Curve (AUC) of Risdiplam | From Day 1 through Day 28
Steady-state Concentration (Css) of Risdiplam | From Day 1 through Day 28
Risdiplam Free Fraction | From Day 1 through Day 28
Percentage of Participants With Adverse Events | Up to 30 days after the final dose of study treatment (up to 58 days)
Percentage of Participants With Serious Adverse Events | Up to 30 days after the final dose of study treatment (up to 58 days)
Percentage of Participants With Treatment Discontinuation due to Adverse Events | Up to 30 days after the final dose of study treatment (up to 58 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (3):
  - Ann and Robert H. Lurie Children Hospital of Chicago, Chicago, Illinois
  - University Of Michigan, Ann Arbor, Michigan
  - Clinic for Special Children., Gordonville, Pennsylvania
- Belgium (2):
  - Hopital Universitaire des Enfants Reine Fabiola, Brussels
  - CHR Citadelle, Liège
- Children'S Hospital of Eastern Ontario, Ottawa, Ontario, Canada
- Universitatsklinikum Essen, Essen, Germany
- Italy (2):
  - Fondazione Serena Onlus - CENTRO CLINICO NEMO, Milano, Emilia-Romagna
  - Fondazione Policlinico Univeristario A. Gemelli, ROMA, Emilia-Romagna
- UMC Utrecht, Utrecht, Netherlands
- OUS (Oslo University Hospital), Rikshospitalet, Oslo, Norway
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing